CLINICAL TRIAL: NCT05780632
Title: A Prospective Observational Study of Biomarkers for a Personalised IVF Treatment,
Brief Title: A Prospective Observational Study of Biomarkers for a Personalised IVF Treatment
Acronym: NAITIVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cognitive IVF a.s. (Other)
Collaborators: Brno University Hospital (Other); Hospital General Universitario Morales Meseguer (Other); Gynem (Unknown); Pronatal (Unknown); Szentagothai research centre (Unknown); University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: LEEAF10032023
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Poor Response to Ovulation Induction
Keywords: ovarian stimulation; IVF; oocyte; environment; algorithm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, follicular fluid, embryonic culture media
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study investigates the effect of four-dimensional patient data (medical, lifestyle, environmental, and genetic) on the outcomes of ovarian stimulation for IVF.

Study will allow us to create a meaningful combination of medical knowledge, unique physician experience and information derived from data analysis. Additionally, the Study allows us to fine-tune the existing algorithms and develop new decision-supporting algorithms.

DETAILED DESCRIPTION:
Details of the ovarian stimulation and its outcomes for each patient will be analysed with the corresponding patient data collected or generated during the Study in the five streams as described under the headings "Stream one" to "Stream five".

Stream one: Personal and medical data Patient mobile app - collects up to 227 different data points about the female and additional up to 64 data points about her partner, Appendix 13.

Physician portal - mirrors the patient data from the mobile app and will provide tools for physician decision-making support and for error minimisation during the treatment using algorithms.

Stream two: Biorhythms and lifestyle Devices monitoring activity and health data (smart watches, bracelets, rings)

1. Heart rate
2. Respiratory rate
3. Heart rate variability
4. Blood oxygen level
5. Sleeping cycle
6. Sleeping respiratory rate
7. Body temperature
8. Activity - steps
9. Stress level

Stream three: Environment

Based on patient location(s), the following data are monitored:

1. Season
2. Weather
3. Moon phases
4. Sun activity
5. Pollution

Stream four: Biomarkers Blood tests - the hormonal profile is determined at the beginning of the menstrual cycle and some determinations are made on the day of ovulation induction (trigger)

1. anti-mullerian hormone
2. follicle stimulating hormone
3. luteinizing hormone (also on the trigger day)
4. Oestradiol (also on the trigger day)
5. Prolactin
6. Progesterone (also on the trigger day)
7. thyroid-stimulating hormone (TSH)
8. antibody thyroid peroxidase
9. sex hormone-binding globulin
10. Testosterone
11. DHEAS

Follicular fluid (FF)

1. Examination of oxidative stress level a. Total oxidant status, Appendix 14 b. Total antioxidant capacity, Appendix 14
2. Proteomic analysis, Appendix 15
3. Amino acids analysis, Appendix 15
4. Lipidaemic analysis, Appendix 15
5. Metabolomic analysis, Appendix 15

Cumulus cells (CCs) a) Telomere length and telomere activity analysis, cell viability score, Appendix 16

Embryonic culture media (ECM)

a) Embryonic DNA analysis by Next Generation Sequencing (NGS), Appendix 17 b) Embryonic microRNA analysis, Appendix 17 Stream five: Genetic study of FSH-receptor and polycystic ovary syndrome polymorphisms

1. Polymorphisms of gene receptors influencing the response to ovarian stimulation by Next-Generation Sequencing (NGS) a. follicle-stimulating hormone receptor
2. Gene polymorphisms in polycystic ovary syndrome patients a. CYP11A1 b. CYP17A1 c. CYP19A1

ELIGIBILITY:
Inclusion Criteria:

1. women aged 18-45 accompanied by a male partner;
2. diagnosis of infertility: one year of unprotected intercourse for patients under the age of 35; 6 months for patients aged 35 and older;
3. embryo transfer planned using fresh, autologous oocytes;
4. using the Oura Ring smart device and sharing health and lifestyle data through the device at least during the IVF treatment (from the beginning of ovarian stimulation until the pregnancy test).

Exclusion Criteria:

1. history of cancer or use of chemotherapeutic agents;
2. history of autoimmune disease (apart from thyroid disease);
3. known genetic conditions or balanced translocations causing disease or risk of disease which may require pre-implantation genetic testing;
4. use of donated oocytes;
5. stimulation protocols without polycystic ovary syndrome analogues.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients undergoing IVF treatment
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
number of mature competent oocytes | 24 months
  quality of oocytes which ensures high fertilisation rate

CONTACTS AND LOCATIONS:
Overall Officials: Jan Choma, MS, Principal Investigator — Cognitive IVF
Locations (1):
- Pronatal, Ostrava, Czechia